CLINICAL TRIAL: NCT04959448
Title: Assessing Long-Term Outcomes of DUPIXENT® Treatment in Patients With Chronic Rhinosinusitis With Nasal Polyposis (AROMA)
Brief Title: Study Assessing Long-teRm Outcomes of dupiluMAb (DUPIXENT®) Treatment in Adult Patients With Chronic Rhinosinusitis With Nasal Polyposis (CRSwNP)
Acronym: AROMA
Status: Active, not recruiting | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: R668-cSNP-2072; 42822 (Registry Identifier: EU HMA-EMA Catalogue)
Record Dates: First submitted 2021-06-21; First posted 2021-07-13 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyposis
Keywords: CRSwNP
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: DUPIXENT® — No investigational agents will be provided. All treatments will be prescribed at the discretion of the study physician and other healthcare providers.
  Other Names: dupilumab; REGN668; SAR231893

SUMMARY:
The primary objectives of the study are:

* To longitudinally characterize the long-term effectiveness of DUPIXENT® through assessment of patient-reported symptoms, Health-Related Quality of Life (HRQoL) related to Chronic rhinosinusitis with nasal polyposis (CRSwNP) and other type 2 comorbidities, and their change over-time.
* To characterize patients who receive DUPIXENT® for CRSwNP in a real-world setting with respect to their medical history, demographic and disease characteristics, and type 2 comorbidities

The secondary objectives of the study are:

* To characterize real-world utilization of DUPIXENT® for patients with CRSwNP
* To collect patient and physician global assessment of disease severity and treatment satisfaction for patients receiving DUPIXENT® for CRSwNP
* To collect long-term safety data for patients receiving DUPIXENT® for CRSwNP

ELIGIBILITY:
Key Inclusion Criteria:

* All patients who are newly initiated on DUPIXENT® for the treatment of CRSwNP according to the respective prescribing information (Product Label or SmPC)
* Willing and able to comply with clinic visits and study-related procedures as per protocol
* Provide informed consent signed by study patient or legally acceptable representative
* Able to understand and complete study-related questionnaires as per protocol

Key Exclusion Criteria:

* Patients who have a contraindication to DUPIXENT® according to the country-specific prescribing information
* Any previous treatment with DUPIXENT® for any condition
* Any condition that, in the opinion of the investigator, may interfere with the patient's ability to participate in the study per protocol
* Participation in an ongoing interventional or observational study that might, in the treating physician's opinion, influence the assessments for the current study per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are initiating treatment with DUPIXENT® for CRSwNP according to the country-specific prescribing information.
Sampling Method: Non-Probability Sample
Enrollment: 717 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2027-03-25 (Estimated); Study Completion 2027-03-25 (Estimated)

PRIMARY OUTCOMES:
Baseline Patient Characteristics | Baseline up to 3 years
  Demographics includes but is not limited to gender, age, ethnicity, height, weight, BMI, education, current employment status, physician information.
Baseline Disease Characteristics | Baseline up to 3 years
  Medical History includes but is not limited to history of CRSwNP, comorbid conditions, age at CRSwNP diagnosis, and baseline measurements of effectiveness variables.

SECONDARY OUTCOMES:
DUPIXENT® Treatment Characteristics | Baseline up to 3 years
  Including but not limited to: usage, dosage, adherence, interruption, place (home or clinic) and frequency of administration
CRSwNP Treatment Characteristics | Baseline up to 3 years
  Including but not limited to: usage, dosage, adherence, duration and frequency
Incidence and severity of adverse events (AEs) | Baseline up to 3 years
Participant Assessment: Total symptom score (TSS), including sub-scores (nasal congestion [NC] and loss of smell [LOS]) | Baseline up to 3 years
  The TSS is a composite score (ranging between 0 and 9) and consisting of the sum of the following symptoms assessed daily: nasal congestion/obstruction, decreased/loss of sense of smell, rhinorrhea (average of anterior/posterior nasal discharge). Higher scores indicate greater symptom burden.
Physician Assessment: Change in University of Pennsylvania Smell Identification Test (UPSIT) score | Baseline up to 3 years
  The UPSIT (UPSIT 40-odorant test) is a rapid and easy-to-administer method to quantitatively assess human olfactory function.
Physician Assessment: CT-Lund-Mackay Score | Baseline up to 3 years
  The LMK system is scoring based on CT imaging of the sinuses with points given for degree of opacification:
  0 = no opacification, 1 = partial opacification, 2 = total opacification. These points are then applied to the maxillary, anterior ethmoid, posterior ethmoid, sphenoid, frontal sinus on each side. The ostiomeatal complex is graded as 0 = not occluded, or 2 = occluded. The sum of these derives a maximum score of 12 per side and 24 in total.
Physician Assessment: Nasal Peak Inspiratory Flow (PNIF) | Baseline up to 3 years
  Nasal peak inspiratory flow (NPIF) is a measure of the air flow through both nasal cavities during forced inspiration expressed in liters per minute.
Physician Assessment: - Forced Expiratory Volume in 1 second (FEV1) | Baseline up to 3 years
  Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled in the first second of a forced exhalation
Physician Assessment: Fractional exhaled Nitric Oxide (FeNO) | Baseline up to 3 Years
  FeNO (Fractional exhaled Nitric Oxiide) is analyzed using a respiratory flow rate of 50 mL/second and reported in ppb.
Participant Assessment: Asthma Control Questionnaire, 6-item (ACQ-6) | Baseline up to 3 Years
  The ACQ-6 assesses asthma control with scores ranging from 0 (fully controlled; 6=severely uncontrolled).
Participant Assessment: Mini Asthma Quality of Life Questionnaire (MiniAQLQ) | Baseline up to 3 Years
  The MiniAQLQ is assesses the impact of asthma on health-related quality of life with scores ranging from 1 (maximum impairment) to 7 (no impairment).
Participant Assessment: Allergic Rhinitis (AR) using AR Visual Analog Scale (VAS) | Baseline up to 3 Years
  The AR-VAS assesses severity of rhinosinusitis symptoms on a 0 (not troublesome) to 10 (worst thinkable troublesome) scale.
Participant Assessment: Mini Rhinoconjunctivitis Quality of Life Questionnaire (MiniRQLQ) | Baseline up to 3 Years
  The MiniRQLQ is an abbreviated version of the RQLQ(S)+12 which assesses health-related quality of life associated with perennial or seasonal allergic rhinitis with scores ranging from 0 (not troubled) to 6 (extremely troubled).
Participant Assessment: Sino-Nasal Outcome Test (SNOT-22) | Baseline up to 3 Years
  The SNOT-22 assesses the impact of chronic rhinosinusitis on health-related quality of life with scores ranging from 0 to 110; lower scores representing better health related quality of life.
Participant Assessment: Patient Oriented Eczema Measure (POEM) | Baseline up to 3 Years
  The POEM assesses symptoms of dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping with scores ranging from 0 to 28; higher scores indicate greater symptom burden.
Participant Assessment: Work Productivity and Activity Impairment Questionnaire for asthma (WPAI-CRSwNP) | Baseline up to 3 Years
  The WPAI-CRSwNP measures impairments in work and activities associated with CRSwNP. Scores are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Physician Assessment: Changes of Healthcare Utilization | Baseline up to 3 years
  Resource use collected from medical, hospital, and pharmacy records
Participant Assessment: Short Form 12 | Baseline up to 3 years
  The SF-12 assesses physical functioning, social functioning, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy/vitality, pain, and general health perception with scores ranging from 0 to 100; lower scores represent greater quality of life impairment.
Participant Assessment: European Quality of Life 5-Dimensions, 5-Level Questionnaire (EQ-5D-5L) | Baseline up to 3 years
  The EQ 5D-5L descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and the EQ-VAS records the respondent's self rated health on a scale of 0 (worst imaginable health state) to 100 (best imaginable health state).
Participant Assessment: Global Impression for Symptom Severity, Treatment Satisfaction (Global Patient Assessment) | Baseline up to 3 years
  The Global Patient Assessment is a 2-component questionnaire on symptom severity over the past week and the patient's overall satisfaction with their CRSwNP treatment.
Physician Assessment: Global Impression for Disease Severity (Global Physician Assessment) | Baseline up to 3 years
  The Global Physician Assessment is a 1-item question asking physicians to rate the severity of their patient's CRSwNP.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (81):
- United States (48):
  - Excel ENT of Alabama, Birmingham, Alabama
  - Medical Research of Arizona, a division of Allergy, Asthma & Immunology Associates, Scottsdale, Arizona
  - The Allergy and Rheumatology Medical Clinic, La Jolla, California
  - ARK Clinical Research, Long Beach, California
  - Scripps Health - Scripps Clinic Carmel Valley, San Diego, California
  - Breathe Clear Institute, Torrance, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - AADRS Clincial Research Center, Coral Gables, Florida
  - University of Florida, Gainesville, Florida
  - Damask Physicians Group, Lake Mary, Florida
  - University of South Florida, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - IACT Health, Columbus, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - The University of Chicago Medical Center UCMC Duchossois Center for Advanced Medicine DCAM, Chicago, Illinois
  - Asthma & Allergy Center of Chicago, Oak Park, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - John Hopkins University School Of Medicine, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan, Michigan Medicine Pulmonary Clinic, Ann Arbor, Michigan
  - Allergy & Asthma Center of Minnesota - Allergology, Maplewood, Minnesota
  - University of Missouri, Columbia, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Atlantic Research Center LLC, Ocean City, New Jersey
  - Northwell Health, Great Neck, New York
  - Montefiore Medical Center, New York, New York
  - Rochester Regional Health System, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Allergy Partners of the Triangle, Raleigh, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Essential Medical Research, Tulsa, Oklahoma
  - Asthma, Nasal Disease & Allergy Research Center of New England, East Providence, Rhode Island
  - Allergy and Asthma Physicians of RI, Lincoln, Rhode Island
  - Medical University Of South Carolina, Charleston, South Carolina
  - ADAC research, PA, Greenville, South Carolina
  - Spartanburg Ear, Nose & Throat Clinical, Spartanburg, South Carolina
  - ENT & Allergy Partners, Summerville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - STAAMP Research, San Antonio, Texas
  - Tanner Clinic, Layton, Utah
  - University of Virginia Health System (UVA), Charlottesville, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Richmond Ear Nose & Throat, Richmond, Virginia
  - The Vancouver Clinic, Vancouver, Washington
- Canada (5):
  - ENT Clinic Sinus Center, St. Paul's Hospital, Vancouver, British Columbia
  - Dr. Richard Gall Med Corp, Winnipeg, Manitoba
  - Toronto Allergy & Asthma Clinic-Pulmonology, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Hopital Du Saint-Sacrement, Québec
- Germany (8):
  - University Hospital Mannheim - Dermatology, Venerology, Allergology, Mannheim, Baden-Wurttemberg
  - Charité, Berlin, Brandenburg
  - Oberhavelkliniken Hennigsdorf, Hennigsdorf, Brandenburg
  - Zentrum für Rhinologie, Wiesbaden, Hesse
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - University Hospital Münster, Münster, North Rhine-Westphalia
  - Praxis Dr. Yury Yarin, Dresden, Saxony
  - Universitätsklinikum Jena, Jena, Thuringia
- Italy (10):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliero Universitara Policlinico di Catania, Catania, Sicily
  - Universita Degli Studi di Pisa Ospedale di Cisanello Pisa, Pisa, Tuscany
  - Azienda Ospedaliero Universitaria Senese, Siena, Tuscany
  - AOU di Padova, Padua, Veneto
  - Università Degli Studi Magna Graecia di Catanzaro, Catanzaro
  - ENT Clinic San Martino Hospital, Genova
  - Azienda Policlinico Umberto I - Università degli Studi di Roma "La Sapienza", Rome
  - Fondazione universitaria Policlinico A. Gemelli, Rome
  - Azienda Ospedaliero Universitaria di Sassari, Sassari
- Japan (7):
  - University of Fukui Hospital - Otorhinolaryngology, Yoshida-gun, Hukui
  - Fujisawa City Hospital, Fujisawa, Kanagawa
  - Nagaoka Red Cross Hospital - Otorhinolaryngology, Nagaoka, Niigita
  - Osaka Haibikino Medical Center, Habikino, Osaka
  - Tokyo Kyosai Hospital, Meguro-Ku, Tokyo
  - Matsuwaki Clinic Shinagawa, Shinagawa-Ku, Tokyo
  - Kyoto Nose & Allergy Clinic, Kyoto
- Netherlands (3):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland
  - Amsterdam UMC location AMC, Amsterdam, North Holland
  - Alrijne Ziekenhuis, Leiderdorp, South Holland

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Siddiqui S, Bachert C, Chaker AM, Han JK, Hellings PW, Peters AT, Heffler E, Kamat S, Zhang H, Nash S, Khan AH, De Prado Gomez L, Jacob-Nara JA, Rowe PJ, Deniz Y. AROMA: real-world global registry of dupilumab for chronic rhinosinusitis with nasal polyps. ERJ Open Res. 2022 Nov 28;8(4):00085-2022. doi: 10.1183/23120541.00085-2022. eCollection 2022 Oct. PMID 36451848
- See also: THE AROMA LANDMARK REGISTRY: A GLOBAL STUDY INVOLVING AN APPROVED INJECTABLE MEDICINE FOR CHRONIC RHINOSINUSITIS WITH NASAL POLYPS — https://np-aromastudy.com/